## First Face Healing Lodge Training Evaluation Study: Analytic Plan February 21, 2024

After all data are collected, the investigators will calculate aggregate scores for the primary outcomes on each occasion. The seven primary outcomes will be (1) total First Face knowledge assessment scores, (2-6) **five** subscale mean scores on the Attitudes Towards Serious Mental Illness - Adolescent Version (ATSMI-AV), and (7) mean Perceived Competence to Respond (PCR) scores. They will report internal consistency of the ATSMI-AV subscales and PCR at pre-training. They will create three change scores for each outcome variable: post-training minus pre-training, 3-month minus post-training, and 3-month minus pre-training. The investigators will generate and report descriptive statistics on all measures.

To study the immediate effects of First Face training on the seven primary outcomes, they will use separate ANOVAs on each outcome with time (pre-training, post-training) as the within-subjects factor and 4 participant characteristics (i.e. Healing Lodge department (coded as direct care provider vs. other), Tribal affiliation (coded as yes or no), residence on a reservation (coded as yes or no), and years worked with at-risk children (code as above the median or at/below the median) as between-subjects factors. Cases with missing data will be deleted listwise. They will note any primary outcomes that show a statistically significant main effect of time. Additionally, they will identify each statistically significant interaction between time and a single between-subjects factor. For each statistically significant 2-way interaction between time and a single between-subjects factor, they will decompose the interaction by conducting paired samples Bonferroni-adjusted *t*-tests at each level of the between-subjects factor.

The investigators will then turn to the three secondary outcomes collected at post-training: (1) satisfaction with training (Likert-type scale), (2) intention to use training in one's professional life (4-category scale from "not at all" to "to a great extent"), (3) intention to use training in one's personal life (4-category scale from "not at all" to "to a great extent"). They will use *t*-tests to determine if the 4 between-subject factors (i.e. Healing Lodge department (coded as direct care provider vs. other), Tribal affiliation (coded as yes or no), residence on a reservation (coded as yes or no), and years worked with at-risk children (code as above the median or at/below the median) are related to these secondary outcomes, as cell sizes permit.

When 3-month follow-up data have been collected, the investigators will conduct attrition analyses to determine if 5 participant characteristics (i.e. Healing Lodge department (coded as direct care provider vs. other), Tribal affiliation (coded as yes or no), residence on a reservation (coded as yes or no), and years worked with at-risk children) and satisfaction with training (coded as very dissatisfied to neutral vs. slightly satisfied to very satisfied) are associated with

completing the 3-month post-training survey. They will use chi-square to conduct these analyses and report whether any participant group was less likely than anticipated to complete the 3-month follow-up.

The investigators will then examine the extent to which trainees maintain any favorable training effects over time. They will conduct the same repeated measures ANOVAs as described above, except this time they will include 3 levels of time as the within-subjects factor (pre-training, post-training, 3-month follow-up). They will use the same between-subject factors. For each outcome that shows a statistically significant main effect of time, the investigators will decompose the main effect by conducting paired samples Bonferroni-adjusted *t*-tests (pre-training versus 3-month follow-up; post-training versus 3-month follow-up). They will explore 2-way interactions between time and a single between-subjects factor as described above.

They will examine the three secondary outcomes reported at the 3-month follow-up: opportunity to use the training (yes or no), use of training in one's personal life (yes or no), and barriers to using training (yes or no for each barrier). They will use chi-square to determine if the 4 between-subject factors (i.e. Healing Lodge department (coded as direct care provider vs. other), Tribal affiliation (coded as yes or no), residence on a reservation (coded as yes or no), and years worked with at-risk children (code as above the median or at/below the median) are related to the secondary outcomes, as cell sizes permit.

The investigators will use Pearson correlation or point-biserial correlation to determine if the 7 primary outcomes are related to the secondary outcomes (as cell sizes permit).

The investigators hypothesize that participants will show favorable improvements on all primary outcomes from pre-training to post-training and from pre-training to 3-month follow-up with no observable change from post-training to 3-month follow-up.